CLINICAL TRIAL: NCT00761696
Title: A Phase 1 Study of IPI-926 in Patients With Advanced and/or Metastatic Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-926-01
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Neoplasms
Keywords: solid tumor malignancies
MeSH Terms: conditions — Neoplasms | interventions — IPI-926

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-926 (Experimental): Oral daily dosing
  Interventions: Drug: IPI-926

INTERVENTIONS:
Drug: IPI-926 — Oral daily dosing
  Other Names: Hedgehog pathway inhibitor

SUMMARY:
The primary objectives of the study are:

* To determine the safety and the maximum tolerated dose (MTD) of IPI-926
* To examine the pharmacokinetic parameters of IPI-926 and its characterized major metabolite(s)
* To recommend a dose and schedule of IPI-926 for subsequent studies

DETAILED DESCRIPTION:
Study IPI-926-01 is a Phase 1, open-label, dose-escalation study in patients with advanced and/or metastatic solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of a solid tumor for which no standard therapy proven to provide clinical benefit is available.
2. ≥18 years of age
3. Life expectancy of at least 3 months.
4. ECOG performance status of 0 to 2.
5. Ability to follow the study and all protocol requirements.
6. Voluntarily sign an informed consent form
7. Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation of who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum or urine pregnancy test prior to treatment. All WCBP, all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study.
8. Recovery to </= Grade 1 or baseline of any toxicities due to prior treatments, excluding alopecia.

Exclusion Criteria:

1. Treatment with following therapies as indicated:

   * Any chemotherapy (other than nitrosoureas or mitomycin C), radiation therapy, surgery, hormonal therapy, or investigational therapy within 4 weeks of the start of IPI-926 administration. Patients with luteinizing hormone releasing hormone therapy.
   * Any tyrosine kinase inhibitor (e.g. erlotinib, imatinib) within 2 weeks of the start of IPI-926 administration
   * Nitrosoureas o or mitomycin C within 6 weeks of the start of IPI-926 administration.
2. Inadequate hematologic function - neutrophil count (ANC) <1,500 cells/mm3, platelet count <100,000/mm3, or hemoglobin <9.0 g/dL (may be increased to this level with transfusion as long as there is no evidence of active bleeding).
3. Inadequate hepatic function - aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN); >5 x ULN if attributable to liver metastases; total bilirubin >1.5 x ULN.
4. Inadequate renal function - serum creatinine >1.5 x ULN.
5. Uncontrolled hypomagnesemia or hypokalemia, defined as ≥ Grade 3 despite adequate electrolyte supplementation.
6. Baseline QTcF >450 msec in men or >470 msec in women.
7. Concurrent treatment with any agent known to prolong the QTc interval.
8. Prior surgery affecting drug absorption or any gastrointestinal dysfunction that could alter drug absorption (e.g. gastric bypass, Whipple procedure, gastrectomy).
9. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
10. Venous thromboembolic event (e.g. pulmonary embolism or deep vein thrombosis) requiring anticoagulation or who meet any of the following criteria are excluded:

    * have been on a stable dose of anticoagulation for <1 month
    * have had a Grade 2, 3 or 4 hemorrhage in the last 30 days
    * experiencing continued symptoms from venous thromboembolic event (e.g. continued dyspnea or oxygen requirement) *Past venous thromboembolic event but do not meet any of the above three criteria are eligible for participation.
11. History of a seizure within the last 10 years or seizure disorder requiring anti-epileptic medications.
12. Concurrent treatment with medications known to lower the seizure threshold.
13. Concurrent administration of the medications or foods which are known to inhibit or induce CYP3A activity to a clinically relevant degree.
14. Presence of active infection or systemic use of antibiotics within 72 hours of treatment.
15. Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study.
16. Known immunodeficiency virus (HIV) positivity.
17. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety and the maximum tolerated dose (MTD) of IPI-926 | 6mths to 1 year

SECONDARY OUTCOMES:
To evaluate the anti-tumor activity of IPI-926 | 6mths to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (5):
- United States (4):
  - TGen Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - Stanford University, Redwood City, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - Johns Hopkins Uninversity, Baltimore, Maryland
- McGill University Jewish General Hospital, Montreal, Quebec, Canada